CLINICAL TRIAL: NCT06699706
Title: Neuroimage-guided Dual-target Continuous Theta Burst Stimulation for Generalized Anxiety Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, phD, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-cTBS-anxiety
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Transcranial Magnetic Stimulation Repetitive
Keywords: Transcranial Magnetic Stimulation; anxiety; neuroimage
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active cTBS group (Active Comparator): Dual-target active cTBS will be performed over 7 consecutive days
  Interventions: Other: Continuous theta-burst stimulation
- sham cTBS group (Sham Comparator): Sham stimulation of dual-target cTBS was performed for 7 consecutive days using a sham coil
  Interventions: Other: sham continuous theta-burst stimulation

INTERVENTIONS:
Other: Continuous theta-burst stimulation — cTBS targets two regions: the dorsolateral prefrontal cortex (dlPFC) and the M1 area. Before the first treatment, each participant's resting motor threshold (RMT) will be determined using a five-step procedure for the primary motor cortex. RMT is defined as the minimum intensity required to elicit a motor response greater than 50 µV in at least 5 out of 10 consecutive trials in the right first dorsal interosseous muscle.
  Participants will then undergo daily cTBS treatment three times a day for 7 consecutive days. Each stimulation session lasts 40 seconds, consisting of triplets of 50 Hz theta-burst stimulation repeated at 5 Hz, delivering a total of 600 pulses. Stimulation of the dlPFC target will be immediately followed by stimulation of the M1 target. To achieve cumulative aftereffects, the protocol will be repeated three times per day (a total of 3600 pulses/day) with two 15-minute breaks between sessions, timed with a stopwatch.
  Arms: active cTBS group
Other: sham continuous theta-burst stimulation — The treatment pattern for the sham continuous theta-burst stimulation was similar to that for real stimulation. The sham coil is identical in appearance to the active coil, but it only produces sounds and sensations similar to those of the active coil on the scalp without generating a current, preventing participants from identifying their group assignment.
  Arms: sham cTBS group

SUMMARY:
The aim of this clinical trial was to determine whether image-guided dual-target cTBS is effective for anxiety disorders. The main questions it aims to answer are:

1. Does dual-target cTBS improve patients' anxiety symptoms?
2. Does dual-target cTBS improve patients' somatization symptoms?
3. Researchers will compare cTBS real and sham stimulation to determine whether cTBS is effective in treating anxiety disorders.

Participants will:

1. Received either cTBS treatment or sham stimulation for 7 consecutive days
2. Psychological assessment and MRI scan were performed before treatment, within 2 days, 2 weeks and 1 month after treatment
3. Adverse reactions during the experiment were recorded

DETAILED DESCRIPTION:
This was a randomized, double-blind, sham-controlled clinical trial. Patients with generalized anxiety disorder (GAD) were recruited from the Neurology Outpatient Clinic and Psychiatry Outpatient Clinic at the First Affiliated Hospital of Anhui Medical University, as well as the Psychiatry Outpatient Clinic and Inpatient Ward at the Second Affiliated Hospital of Anhui Medical University. The diagnosis of GAD was based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), independently confirmed by two professional psychiatrists. Patients meeting the inclusion criteria provided written informed consent and were randomly assigned to either a true cTBS treatment group or a sham stimulation group.

Patients will be randomly assigned to receive either active or sham cTBS treatments according to a computer-generated list by an unblinded investigator not involved with study ratings/analysis. The assignment will be executed by utilizing sealed opaque envelopes, each containing the code corresponding to the assigned group for every participant. To ensure the integrity of the double-blind procedure, patients, clinical raters, and all personnel responsible for the clinical care of patients will remain uninformed about the assigned condition until the end point of study. Only cTBS administrators have access to the randomization list. The patients, clinical assessors, and all personnel responsible for clinical care remained blinded to group allocation.

After randomization, patients underwent 7 days of cTBS treatment and completed psychological evaluations and multimodal MRI scans at three time points: baseline, post-treatment, and follow-up. Baseline evaluations were conducted within 24 hours before the first cTBS session, while post-treatment and follow-up evaluations were performed 24 hours after the final cTBS session and four weeks later, respectively.

At each time point (baseline, post-treatment, and follow-up), trained evaluators conducted MRI scans and administered the following scales and behavioral paradigms:

Hamilton Anxiety Rating Scale (HAMA); Hamilton Depression Rating Scale (HAMD); Patient Health Questionnaire-15 (PHQ-15); Self-Rating Anxiety Scale (SAS); Insomnia Severity Index (ISI); MFTM-A (Cognitive Control Capacity); Attention Network Test (ANT).

These scales and paradigms were used to assess the severity of symptoms across different dimensions of anxiety. Additionally, demographic data, structural MRI (sMRI), and functional MRI (fMRI) data were collected at baseline. The sMRI data were utilized for real-time navigation during stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. the patients were diagnosed by more than 2 psychiatrists and met the diagnostic criteria of DSM-5 for anxiety
2. HAMA score ≥ 14 (HAMD score < 17).
3. Age range: 18-60 years.
4. Right-handed.
5. Able to cooperate with the collection of general demographic information and neuropsychological testing.
6. Patients are either medication-free or maintain a consistent medication regimen during cTBS treatment.-

Exclusion Criteria:

1. Presence of organic brain lesions detected on MRI.
2. History of alcohol or drug dependence.
3. Diagnosis of other neuropsychiatric disorders, such as epilepsy, autism, obsessive-compulsive disorder, or autoimmune encephalitis.
4. Contraindications to MRI scanning.-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAMA) | 0week, 1week, 3week, 5week
  the change of anxiety symptoms assessed by HAMA scale(Hamilton Anxiety Scale) will constitute the major research outcome measure, to assess response to tACS. HAMA scale scores range from 0 to 56 points, the higher the score indicates the more serious anxiety symptoms

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | 0week, 1week, 3week, 5week
  The Hamilton Depression Rating Scale (HAMD) is a widely-used clinician-rated tool for assessing depression severity. It evaluates mood, physical, and cognitive symptoms through 17-24 items scored 0-2 or 0-4, with total scores categorizing severity from normal (≤7) to severe (≥24).
Patient Health Questionnaire (PHQ-15) | 0week, 1week
  the change of somatic symptoms will be assessed by Patient Health Questionnaire (PHQ-15). PHQ-15 is composed of 15 physical symptoms that have been extracted from the PHQ. PHQ-15 scale scores range from 0 to 30 points. Higher scores indicate more severe somatic symptoms.
Self-rating anxiety scale(SAS) | 0week, 1week
  Self-rating anxiety scale(SAS) is a supplementary evaluation of the change of anxiety state of patients in this experiment, and it also belongs to the category of self-rating scale. Patients assessed anxiety by checking the frequency of 20 items: none or almost none, sometimes, most of the time, most of the time, or all of the time. SAS scale scores range from 0 to 100 points。The higher the score, the more serious the anxiety symptoms.
ISI(The insomnia severity index) | 0week, 1week
  ISI(The insomnia severity index) is used to evaluate the changes of sleep status of anxiety patients in the recent (2 weeks), which is a self-rating scale. ISI scale scores range from 0 to 28 points. The higher the score is, the worse the sleep quality is. This scale indirectly reflects the changes of patients' anxiety state through evaluation.
Attention Network Test (ANT) | 0week, 1week
  The Attention Network Test (ANT) is a computerized cognitive task designed to measure the efficiency of three distinct attention networks:
  Alerting - The ability to achieve and maintain an alert state (measured by the benefit of cueing).
  Orienting - The ability to selectively focus attention (measured by spatial cueing effects).
  Executive Control - The ability to resolve conflict (measured by flanker interference effects).
  Participants respond to a central target stimulus (e.g., an arrow direction) while ignoring distractors (flanker arrows). Reaction time differences between onditions quantify each network's efficiency. The ANT is widely used in cognitive neuroscience and clinical research to study attention deficits in disorders like ADHD, anxiety, and dementia.
MFTM-A (Cognitive Control Capacity) | 0week, 1week
  The MFTM-A (Mental Flexibility Task Module - Adaptive) is a computerized cognitive test measuring executive control capacity, particularly mental flexibility. Using adaptive rule-switching tasks, it assesses:Switch costs (performance differences between rule shifts); Adaptive thresholds (max difficulty achieved); Error monitoring (correction rates). Widely applied in psychiatric research, it offers automated, sensitive evaluation of cognitive flexibility deficits.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No